CLINICAL TRIAL: NCT01881152
Title: Cluster Randomized Controlled Trial to Assess the Effectiveness of a Population-based Educational Campaign on Stroke Symptom Recognition in Reducing Pre-hospital Delay
Brief Title: Effectiveness of a Public Campaign to Increase Stroke Awareness in Reducing Prehospital Delay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Licia Denti, Medical Doctor, Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRUa2-2010-013
Record Dates: First submitted 2013-06-07; First posted 2013-06-19 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Acute Stroke
Keywords: Stroke; Community education; Awareness; Prehospital delay
MeSH Terms: conditions — Stroke; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Educational campaign
  Interventions: Other: Educational campaign
- Control (Other): Usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Educational campaign — Multilevel educational campaign on stroke sympton recognition and the need for calling the Emergency Services
  Other Names: Community campaign; Public campaign
  Arms: Intervention
Other: Usual care — Information on stroke usually delivered at the community level.
  Arms: Control

SUMMARY:
The starting hypothesis is that a multilevel educational campaign, specifically developed for the local community, can increase public stroke awareness and reduce pre-hospital delay.

The effectiveness of such intervention will be evaluated according to a cluster randomized, stepped wedged design. The clusters are the four communities of the Area Vasta Emilia Nord, AVEN (Parma, Piacenza, Modena e Reggio Emilia). As analysis Units, we will consider the patients consecutively admitted to the six participating hospitals throughout the study period, for suspected stroke or transitory ischemic attack (TIA).

DETAILED DESCRIPTION:
After a baseline 3 month period, the educational campaign will be sequentially launched in the four communities over four 3 month periods, according to a computer-generated list. The comparison will be the"usual care".

Primary outcome measures: The proportion of patients arriving at the Emergency Department (ED) with suspected stroke or TIA within two hours.

Secondary outcome measures: the proportion of patients with confirmed stroke or TIA diagnosis; the proportion of ischemic stroke patients evaluated for recominanat Tissue Plasminogen Activator (rTPA) therapy; the proportion of patients treated with rTPA; time interval between arrival at the ED and CT scan; for patients treated with rTPA, time interval between arrival at the ED and therapy initiation (door to needle time); death and disability (assessed as modified Rankin Score 3-5) at 1 and 3 month from stroke onset.

ELIGIBILITY:
Inclusion Criteria:

* Patients consecutively admitted to the six participating hospitals for suspected stroke or transitory ischemic attack (TIA), defined as abrupt onset of focal or generalized neurologic deficit of vascular origin.

Exclusion Criteria:

* No information available on the time of stroke onset.
* No informed consent from patient or caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1772 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percentage of early admission | Time interval from stroke onset to arrival at the Emergency Department
  Proportion of patients arriving to the Emergency Department with suspected stroke or TIA within two hours

SECONDARY OUTCOMES:
Poor outcome at 1 month | 1 month from stroke onset
  Death or disability (modified Rankin Scale 3-6)at 1 month
Poor outcome at 3 months | 3 months from stroke onset
  Death or disability (modified Rankin Scale 3-6) at 3 months
Rate of thrombolysis | Up to 4 hours and 30 minutes from stroke onset
  Proportion of patients given thrombolysis
Rate of thrombolysis activation | Up to 3 hours from stroke onset
  Proportion of patients evaluated for thrombolysis
Delay in CT scan | Up to 12 hours from admission at the ED
  Time interval between arrival at the Emergency Department and CT scan
Door to needle time | Up to 4 hours and 30 minutes from stroke onset
  Time interval between arrival at the ED and thrombolysis initiation

CONTACTS AND LOCATIONS:
Overall Officials: Licia Denti, MD, Principal Investigator — Parma University Hospital
Locations (5):
- Italy (5):
  - AUSL Parma, Fidenza
  - Ospedale Civile S. Agostino Estense-Baggiovara-AUSL Modena, Modena
  - University Hospital of Parma, Parma
  - Ospedale Guglielmo di Siliceto-AUSL Piacenza, Piacenza
  - Arcispedale Santa Maria Nuova of Reggio Emilia, Reggio Emilia

REFERENCES:
- [Derived] Denti L, Caminiti C, Scoditti U, Zini A, Malferrari G, Zedde ML, Guidetti D, Baratti M, Vaghi L, Montanari E, Marcomini B, Riva S, Iezzi E, Castellini P, Olivato S, Barbi F, Perticaroli E, Monaco D, Iafelice I, Bigliardi G, Vandelli L, Guareschi A, Artoni A, Zanferrari C, Schulz PJ. Impact on Prehospital Delay of a Stroke Preparedness Campaign: A SW-RCT (Stepped-Wedge Cluster Randomized Controlled Trial). Stroke. 2017 Dec;48(12):3316-3322. doi: 10.1161/STROKEAHA.117.018135. Epub 2017 Nov 3. PMID 29101258
- [Derived] Caminiti C, Schulz P, Marcomini B, Iezzi E, Riva S, Scoditti U, Zini A, Malferrari G, Zedde ML, Guidetti D, Montanari E, Baratti M, Denti L; Educazione e Ritardo di Ospedalizzazione (E.R.O.I) study group. Development of an education campaign to reduce delays in pre-hospital response to stroke. BMC Emerg Med. 2017 Jun 24;17(1):20. doi: 10.1186/s12873-017-0130-9. PMID 28646851